CLINICAL TRIAL: NCT06441006
Title: Program for Rifampicin-Resistant Disease With Stratified Medicine for Tuberculosis (PRISM-TB)
Brief Title: Program for Rifampicin-Resistant Disease With Stratified Medicine for Tuberculosis
Acronym: PRISM-TB
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7200AA22CA00005; 7200AA22CA00005 (Other Grant/Funding Number: United States Department of State)
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis, MDR
Keywords: Tuberculosis; BPaLM; Bedaquiline; Pretomanid; Linezolid; Moxifloxacin
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis | interventions — bedaquiline; Linezolid; pretomanid; Moxifloxacin

STUDY DESIGN:
Masking Description: PRISM-TB will not include any placebo. Participants, providers, and pharmacists will be aware of strategy and treatment allocation. Masking of participants to treatment allocation would obscure differences in durations and affect behavior in shortened regimens that would not be reflective of future use and is therefore not included as a feature of this trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Strategy 1: Control regimen for all with FQ-S MDR/RR-TB (Active Comparator): The local SOC regimen consistent with preferred regimen(s) in international guidelines. In most cases this will be 24 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (6BPaLM). Doses and durations of each component may change based on the latest international guidelines and the local SOC.
  Interventions: Drug: Control Arm FQ-S MDR/RR-TB regimen, designed according to latest international guidelines
- Strategy 2: 4BPaLM for all with FQ-S MDR/RR-TB (Experimental): 17 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (4BPaLM). Bedaquiline 400 mg orally once daily for 2 weeks, then 200 mg once daily; pretomanid 200 mg orally once daily; linezolid 600 mg orally once daily; and moxifloxacin 400 mg orally once daily.
  Interventions: Drug: Bedaquiline; Drug: Linezolid; Drug: Pretomanid; Drug: Moxifloxacin
- Strategy 3: 3BPaLM or 6BPaLM stratified medicine strategy for those with FQ-S MDR/RR-TB (Experimental): 13 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (3BPaLM) for participants classified as having easier-to-treat TB and 24 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (6BPaLM) for participants classified as having harder-to-treat TB.
  3BPaLM: 13 weeks of bedaquiline 400 mg orally once daily for 2 weeks, then 200 mg once daily; pretomanid 200 mg orally once daily, linezolid 600 mg orally once daily, and moxifloxacin 400 mg orally once daily.
  6BPaLM: 24 weeks of bedaquiline 400 mg orally once daily for 2 weeks, then 200 mg once daily; pretomanid 200 mg orally once daily, linezolid 600 mg orally once daily, and moxifloxacin 400 mg orally once daily.
  Interventions: Drug: Bedaquiline; Drug: Linezolid; Drug: Pretomanid; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Bedaquiline — Frequency: daily Route of administration: oral
  Other Names: Sirturo
  Arms: Strategy 2: 4BPaLM for all with FQ-S MDR/RR-TB; Strategy 3: 3BPaLM or 6BPaLM stratified medicine strategy for those with FQ-S MDR/RR-TB
Drug: Linezolid — Frequency: daily Route of administration: oral
  Other Names: Zyvox
  Arms: Strategy 2: 4BPaLM for all with FQ-S MDR/RR-TB; Strategy 3: 3BPaLM or 6BPaLM stratified medicine strategy for those with FQ-S MDR/RR-TB
Drug: Pretomanid — Frequency: daily Route of administration: oral
  Other Names: Pretamyl
  Arms: Strategy 2: 4BPaLM for all with FQ-S MDR/RR-TB; Strategy 3: 3BPaLM or 6BPaLM stratified medicine strategy for those with FQ-S MDR/RR-TB
Drug: Moxifloxacin — Frequency: daily Route of administration: oral
  Other Names: Avelox
  Arms: Strategy 2: 4BPaLM for all with FQ-S MDR/RR-TB; Strategy 3: 3BPaLM or 6BPaLM stratified medicine strategy for those with FQ-S MDR/RR-TB
Drug: Control Arm FQ-S MDR/RR-TB regimen, designed according to latest international guidelines — The local SOC regimen consistent with preferred regimen(s) in international guidelines. In most cases this will be 24 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (6BPaLM). Doses and durations of each component may change based on the latest international guidelines and the local SOC.
  Arms: Strategy 1: Control regimen for all with FQ-S MDR/RR-TB

SUMMARY:
PRISM-TB is an international, seamless, multicenter, open-label, randomized, controlled, pragmatic, stratified medicine, treatment shortening, multi-arm multi-stage (MAMS), noninferiority Phase 2/3 clinical trial for fluoroquinolone-susceptible multidrug-resistant/rifampin-resistant pulmonary tuberculosis (FQ-S MDR/RR-TB). In Stage 1, participants will be randomized among one of three treatment arms (one control and two experimental). Following the interim analysis (at the end of Stage 1) based on DOOR outcome comparisons and the entirety of the data, one of the four possible experimental strategies will be identified and continue into Stage 2. In Stage 2, participants will be randomized among one of two treatment arms (one control and one experimental).

The trial objective is to identify, among participants with fluoroquinolone-susceptible multidrug-resistant/rifampicin-resistant tuberculosis (FQ-S MDR/RR-TB), the preferred BPaLM strategy of 13 or 17 weeks for participants stratified to receive shorter treatment and 17 or 24 weeks for participants stratified to receive longer treatment, as defined by a prespecified stratification algorithm, and to evaluate whether this BPaLM strategy has noninferior efficacy to the control strategy at Week 73.

DETAILED DESCRIPTION:
At least 200 participants across three treatment arms (67 in each arm) will be enrolled in Stage 1 and at least an additional 200 participants across two treatment arms (100 in each arm) will be enrolled in Stage 2.

Stage 1: After written informed consent, participants with FQ-S MDR/RR-TB will be randomly assigned to receive one of Stage 1 Strategies 1-3.

Stage 1 Strategy 1 (control strategy): Control regimen for all with FQ-S MDR/RR-TB. The local standard of care (SOC) regimen consistent with preferred regimen(s) in international guidelines. In most cases this will be 24 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (6BPaLM). Doses and durations of each component may change based on the latest international guidelines and the local SOC.

Stage 1 Strategy 2 (investigational strategy): 4BPaLM for all with FQ-S MDR/RR-TB. 17 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (4BPaLM).

Stage 1 Strategy 3 (investigational strategy): 3BPaLM or 6BPaLM stratified medicine strategy for FQ-S MDR/RR-TB. 13 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (3BPaLM) for participants stratified to receive shorter treatment and 24 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (6BPaLM) for participants stratified to receive longer treatment.

Stage 2: After written informed consent, participants with FQ-S MDR/RR-TB will be randomly assigned to receive one of the Stage 2 Strategies 1-2.

Stage 2 Strategy 1 (control strategy): Control regimen for all with FQ-S MDR/RR-TB. The local standard of care (SOC) regimen consistent with preferred regimen(s) in international guidelines. In most cases this will be 24 weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (6BPaLM). Doses and durations of each component may change based on the latest international guidelines and the local SOC.

Stage 2 Strategy 2 (investigational strategy): Preferred strategy from Stage 1 for FQ-S MDR/RR-TB. Number of weeks of bedaquiline, pretomanid, linezolid, and moxifloxacin (BPaLM) for participants stratified to receive shorter treatment and for participants stratified to receive longer treatment to be determined from the preferred strategy identified in Stage 1.

The sites listed below are the planned sites for Stage 1 and/or Stage 2.

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all of the following inclusion criteria at the time of enrollment in order to participate in this study:

1. Confirmed fluoroquinolone-susceptible rifampicin-resistant pulmonary tuberculosis, based on sputum Xpert MTB/RIF and Xpert MTB/XDR, and/or other validated molecular test, and/or phenotypic drug susceptibility testing.

   a. NOTE: TB diagnosis for purposes of meeting this inclusion criterion can be from a study testing laboratory or from an outside laboratory.
2. Aged ≥ 14 years.
3. A verifiable address or residence location that is readily available for visiting, willingness to consent to home visits and phone calls, and willingness to inform the study team of any change of address during the treatment and follow-up period.
4. Ability and willingness of individual to provide written informed consent or written consent from a parent, guardian, or caregiver and assent of the child participant per local ethics committee guidance.
5. Documentation of negative HIV infection status within 30 days prior to study entry or documentation confirming HIV infection at any time before study entry.
6. For individuals with HIV: CD4+ cell count ≥ 50 cells/mm3 based on testing performed within 30 days prior to study entry.
7. For individuals with HIV: Currently being treated with dolutegravir-based antiretroviral therapy (ART), or plan to initiate dolutegravir-based ART at or before study week 8.

   a. NOTE: Dosing of ART and chemoprophylaxis for opportunistic infections should be reflective of local standard of care based on WHO or national guidelines. The following antiretrovirals are disallowed given significant drug-drug interactions with bedaquiline: efavirenz, etravirine, all protease inhibitors, and cobicistat-boosted elvitegravir. The following antiretroviral is disallowed given risk of myelosuppression with linezolid: zidovudine.
8. For individuals who are pregnant: at screening, evidence by ultrasound of a viable singleton pregnancy with an estimated gestational age at enrollment of ≥ 14 weeks as per screening ultrasound.
9. Chest radiograph obtained within 14 days prior to study entry.

Exclusion Criteria:

An individual meeting any of the following exclusion criteria at the time of enrollment or initiation of study drugs will be excluded from study participation:

1. Known allergy/sensitivity, intolerance, or any hypersensitivity to components of study TB drugs or their formulation.
2. One or more of the following laboratory parameters:

   1. Absolute neutrophil count (ANC) < 1000/mm3.
   2. Hemoglobin level < 8.0 g/dL.
   3. Serum or plasma alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times the upper limit of normal.
   4. Serum or plasma total bilirubin ≥ 3 times the upper limit of normal.
   5. Serum or plasma creatinine level ≥ 3 times the upper limit of normal.
   6. Evidence of laboratory values consistent with or equivalent to grade 4 toxicity (i.e., potentially life-threatening).
   7. NOTE: Persons found not to be eligible due to laboratory abnormalities may be reevaluated within the screening window.
3. QTcF interval ≥ 480 ms within 5 days prior to study entry.
4. One or more risk factors for QT prolongation (apart from age and sex) or other uncorrected risk factors for torsades de pointes: evidence of ventricular pre-excitation (Wolff-Parkinson-White syndrome); electrocardiographic evidence of either complete left bundle branch block or right bundle branch block, or incomplete left bundle branch block or right bundle branch block and QRS complex duration ≥ 120 ms on at least one ECG; current pacemaker implant; congestive heart failure; evidence of second- or third-degree heart block; bradycardia defined by sinus rate less than 50 bpm; personal or family history of long QT syndrome; personal history of arrhythmic cardiac disease, with the exception of sinus arrhythmia; personal history of syncope (i.e., cardiac syncope not including syncope due to vasovagal or epileptic causes).
5. Current grade 2 or higher peripheral neuropathy.

   a. NOTE: Peripheral neuropathy assessment must be obtained within 7 days prior to study entry.
6. Documentation of Karnofsky Performance Status Score < 50 obtained within 14 days prior to study entry.
7. Known resistance to bedaquiline, pretomanid, delamanid, linezolid, or fluoroquinolones.
8. Previous use of any second-line anti-TB drugs for more than 14 days during the 12 months prior to the screening visit date.
9. Known or presumed central nervous system TB, osteoarticular TB, or miliary/disseminated TB in the current TB episode.
10. Taking any medication that is contraindicated with study medicines which cannot be stopped (with or without replacement) or requires a washout period longer than 2 weeks.
11. Any condition (social or medical or psychological) which, in the opinion of the investigator, would make participation unsafe or interfere with adherence to study requirements.
12. Current enrollment in other therapeutic trials will not be eligible. a. NOTE: Current enrollment of index cases in prevention trials will be allowed on a case-by-case basis, provided that the prevention trial does not include a therapeutic intervention that could affect response to TB treatment.

All persons who are not eligible for the PRISM-TB trial will be managed according to local routine practice and may enroll in other studies.

Criteria for Exclusion after Entry ('Late Exclusion'):

Enrolled individuals who are subsequently determined to meet the following criteria will be classified as 'late exclusions' and study treatment will be discontinued:

1. Bedaquiline, pretomanid, delamanid, linezolid, or fluoroquinolone resistance on phenotypic or molecular drug- susceptibility testing from samples collected up to 4 weeks after randomization.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Outcome: Desirability of Outcome Ranking (DOOR) | 73 weeks
  Desirability of outcome ranking (DOOR) outcome combining efficacy at the end of follow-up (a minimum of 28 weeks post-randomization) and safety at 28 weeks post-randomization.
  DOOR outcomes do not aggregate measures, but rather create distinct ordinal categories that participants will fall under.
  DOOR ordinal categories are as follows:
  1. Cured or treatment completed by end of follow-up and no Grade 3+ AEs and treatment changes;
  2. Cured or treatment completed by end of follow-up and no Grade 3+ with treatment change for any reason;
  3. Cured or treatment completed by end of follow-up and at least one Grade 3+ AE;
  4. Treatment failure or recurrence by end of follow-up and no Grade 3+ AE;
  5. Treatment failure or recurrence by end of follow-up and at least one Grade 3+ AE;
  6. Death by end of follow-up.

SECONDARY OUTCOMES:
Mortality | 73 weeks
  Mortality
All Grade 3 or Higher AEs up to 28 Weeks | 28 weeks
  All Grade 3 or higher AEs up to 28 weeks post-randomization.
All AESIs up to 28 Weeks | 28 weeks
  All AESIs up to 28 weeks post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo E Velásquez, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (6):
- National Center for Communicable Diseases, Ulaanbaatar, Mongolia
- Institute of Chest Diseases, Kotri, Pakistan
- Peru (2):
  - Hospital Nacional Sergio E. Bernales, Lima
  - Policlínico SES, Lima
- Mulago National Referral Hospital, Kampala, Uganda
- Hanoi Lung Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No